CLINICAL TRIAL: NCT01263886
Title: A Multinational, Randomized, Double Blind, Controlled Phase II Trial of Ombrabulin With Taxane and Platinum Combination Administered Every Three Weeks, in First Line Treatment of Patients Metastatic Non-small Cell Lung Cancer
Brief Title: Trial of Ombrabulin (AVE8062) in Combination With Taxane and Platinum in Patients With Non-small Cell Lung Cancer
Acronym: DISRUPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC10259; 2010-019384-11 (EudraCT Number); U1111-1115-3677 (Other: UTN)
Record Dates: First submitted 2010-12-14; First posted 2010-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — AC 7700

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AVE8062 and combination (Experimental): Day 1: AVE8062
  Day 2: docetaxel followed by cisplatin or paclitaxel followed by carboplatin
  Interventions: Drug: ombrabulin (AVE8062)
- Placebo (Placebo Comparator): Day 1: placebo
  Day 2: docetaxel followed by cisplatin or paclitaxel followed by carboplatin
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ombrabulin (AVE8062) — Pharmaceutical form:solution
  Route of administration: intravenous
  Arms: AVE8062 and combination
Drug: placebo — Pharmaceutical form:solution
  Route of administration: intravenous
  Arms: Placebo

SUMMARY:
Primary Objective:

* To demonstrate progression free survival (PFS) improvement for ombrabulin compared to placebo, in combination with taxane and platinum, as first line treatment for patients with metastatic non-small cell lung cancer (NSCLC).

Secondary Objective:

* To determine overall survival (OS), overall response rate (ORR) according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria, safety, and evaluate potential biomarkers, pharmacokinetic (PK) analysis of ombrabulin and its main metabolite, RPR258063, using a population approach.

DETAILED DESCRIPTION:
Patients will be treated for a maximum of 6 cycles (21 days each), in the absence of unacceptable toxicity or disease progression or consent withdrawal. All patients will be followed for disease progression documentation and for patient status until up to one year after the primary analysis cutoff date.

ELIGIBILITY:
Inclusion criteria:

* Histologically proven squamous metastatic non-small cell lung cancer (stage IV, according to Tumor Nodes Metastasis (TNM) classification seventh edition)
* Patients with measurable disease, Response Evaluation Criteria In Solid Tumors (RECIST) criteria (version 1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion criteria:

* Prior chemotherapy, immunotherapy or targeted therapy for lung cancer disease (including adjuvant/neoadjuvant therapy)
* History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis
* History of another neoplasm. Adequately treated basal cell or squamous skin cancer, or in situ cervical cancer, or any other cancer from which the patient has been disease-free for >5 years are allowed
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to randomization
* Acquired immunodeficiency syndrome (AIDS-related illness) or known human immunodeficiency virus (HIV) disease requiring antiretroviral treatment
* Any severe acute or chronic medical condition, which could impair the ability of the patient to participate in the study or interfere with interpretation of study results
* Pregnant or breast-feeding woman. Positive serum or urine pregnancy test prior to randomization
* Patient with reproductive potential (Male/Female) who do not agree to use accepted and effective method of contraception during the study treatment period and for at least 3 months after the completion of the study treatment. The definition of "effective method of contraception" will be based on the investigator's judgment
* Inadequate organ function
* Pre-existing peripheral neuropathy > grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V.4.03
* Pre-existing hearing impairment > grade 2
* Known hypersensitivity due to taxanes and /or polysorbate 80 or any other compound of the study drug combination
* Other serious illness or medical conditions such as (but not restricted): Active infection, Superior vena cava syndrome, Pericardial effusion requiring intervention (drainage)
* Documented medical history of myocardial infarction, documented angina pectoris, arrhythmia especially severe conduction disorder such as second or third-degree atrioventricular block, stroke, or history of arterial or venous thromboembolism within the past 6 months still requiring anticoagulants.
* Uncontrolled hypertension within 3 months prior to study treatment or patient with organ damage related to hypertension.
* Patient with Left Ventricular Ejection Fraction (LVEF) value lower than institution inferior normal limit, evaluated by echocardiography or angiocardiography
* 12-lead Electrocardiogram (ECG): Infarction Q-wave, ST segment depression or elevation ≥1 mm in at least 2 contiguous leads
* History of gross hemoptysis (i.e. 1/2 teaspoon of red blood or more per episode) within the past 1 month.
* Has non-squamous NSCLC(adenocarcinoma/large cell or other)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | approximately 1.5 years

SECONDARY OUTCOMES:
Overall survival (OS) | approximately 1.5 years
Objective response rate (OR) | approximately 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (43):
- United States (5):
  - Investigational Site Number 840001, Muscle Shoals, Alabama
  - Investigational Site Number 840003, Hot Springs, Arkansas
  - Investigational Site Number 840002, Anaheim, California
  - Investigational Site Number 840009, Modesto, California
  - Investigational Site Number 840005, Lansing, Michigan
- Australia (2):
  - Investigational Site Number 036002, Bendigo
  - Investigational Site Number 036001, Southport
- Chile (4):
  - Investigational Site Number 152005, Santiago
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152003, Santiago
  - Investigational Site Number 152004, Valparaíso
- Croatia (3):
  - Investigational Site Number 191002, Zagreb
  - Investigational Site Number 191003, Zagreb
  - Investigational Site Number 191001, Zagreb
- France (5):
  - Investigational Site Number 250005, Bordeaux
  - Investigational Site Number 250002, Dijon
  - Investigational Site Number 250003, Lyon
  - Investigational Site Number 250004, Nice
  - Investigational Site Number 250001, Saint-Herblain
- Germany (3):
  - Investigational Site Number 276001, Gauting
  - Investigational Site Number 276002, Großhansdorf
  - Investigational Site Number 276003, Immenhausen
- Italy (3):
  - Investigational Site Number 380002, Genova
  - Investigational Site Number 380003, Milan
  - Investigational Site Number 380001, Monza
- Poland (4):
  - Investigational Site Number 616003, Lublin
  - Investigational Site Number 616001, Poznan
  - Investigational Site Number 616004, Warsaw
  - Investigational Site Number 616005, Warsaw
- Romania (4):
  - Investigational Site Number 642002, Bucharest
  - Investigational Site Number 642003, Cluj-Napoca
  - Investigational Site Number 642004, Craiova
  - Investigational Site Number 642001, Iași
- Russia (2):
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643004, Saint Petersburg
- Serbia (2):
  - Investigational Site Number 688003, Belgrade
  - Investigational Site Number 688001, Kamenitz
- South Korea (3):
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410002, Seoul
  - Investigational Site Number 410001, Seoul
- Ukraine (3):
  - Investigational Site Number 804001, Dnipropetrovsk
  - Investigational Site Number 804003, Kyiv
  - Investigational Site Number 804002, Sumy